CLINICAL TRIAL: NCT02911740
Title: Investigating the Additive Benefit of the Urine Lipoarabinomannan Test to Current TB Diagnostics Among HIV+ Adults in Panama City, Panama
Brief Title: Additive Benefit of the Urine LAM Test to Current TB Diagnostics in HIV Positive Adults in Panama City, Panama
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Not IRB approved
Sponsor: University of Florida (Other)
Collaborators: Hospital Santo Tomas (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: IRB201600869
Record Dates: First submitted 2016-07-21; First posted 2016-09-22 (Estimated); Last update posted 2017-12-26 (Actual); Status verified 2017-12

CONDITIONS: Tuberculosis; HIV; Histoplasmosis
MeSH Terms: conditions — Tuberculosis; Histoplasmosis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Urine LAM Ag test (Experimental): Patients will be enrolled prospectively and tested for TB using the urine LAM Ag test
  Interventions: Other: Urine LAM Ag test
- Retrospective arm (No Intervention): Charts of retrospectively selected patients from the Hospital Santo Tomas database who presented within the last five years meeting inclusion criteria will be used as controls

INTERVENTIONS:
Other: Urine LAM Ag test — TB diagnostic assay
  Arms: Urine LAM Ag test

SUMMARY:
Tuberculosis (TB) is one opportunistic infection often seen in HIV individuals. In 2013, there were an estimated 31,800 HIV-TB co-infection cases and 6,100 HIV-related deaths due to TB in the Americas. Due to the non-specific nature of its clinical symptoms, TB can be confused with various diseases such as histoplasmosis, sarcoidosis, lymphoma, and pneumonia. In Panama, where Histoplasma capsulatum is endemic, diagnosing TB versus histoplasmosis based on clinical symptoms can be difficult. In Panama, approximately 7.65% of HIV patients are co-infected with histoplasmosis, and there is a 30% mortality rate in HIV-histoplasmosis patients in Latin America. Due to similar clinical features, misdiagnosis of active TB and disseminated histoplasmosis in endemic regions may lead to incorrect antibiotic management, which in turn results in unnecessary toxicity, antibiotic resistance, and monetary expenditures. The investigators interests lie in increasing TB diagnostic accuracy using a simple urine dipstick test and evaluating physician response to new diagnostic testing, in order to reduce misdiagnosis and improve health outcomes in the HIV population.

DETAILED DESCRIPTION:
The gold standard for TB diagnosis, mycobacterial culture, is limited by a slow turnaround time, the need for skilled technicians and biosafety level 3 facilities. Another diagnostic test, Xpert MTB/RIF, produces same-day results, boasts a specificity of 98%, but is limited in the HIV population by its sensitivity of 67% (with a single sputum sample). High costs associated with this test have presented a major obstacle to its routine use (US$65,500 for a 16-module instrument, and US$9.98 to US$18.00 per cartridge). The urine lipoarabinomannan (LAM) Ag test has a specificity of 98.6% and a sensitivity of 66.7% in patients with a CD4 count below 50. LAM is a 17.5kD glycolipid and virulence factor of mycobacteria. The test's sensitivity improves in advanced HIV cases because of the higher bacillary burden, more frequent disseminated TB, and greater concentration of urine antigen due to less antigen-antibody formation, and HIV nephropathy. The test strip contains its own positive and negative controls for quality assurance, and can utilize fresh urine samples stored at room temperature for up to 8 hours after collection. In the right clinical setting, the urine LAM Ag test could have an important additive benefit in TB diagnosis in HIV individuals when combined with the current standards of care.

This study is investigating how physician management and patient outcomes change when the urine LAM test is added to the current TB diagnostic tests (mycobacterial cultures and occasional use of Xpert MTB/RIF). The national referral hospital in Panama, Hospital Santo Tomás, is an ideal study site given its dedicated HIV inpatient service and high TB and histoplasmosis burden. Histoplasmosis diagnosis is often based on clinical symptoms alone, and less frequently confirmed by skin or bone marrow biopsy. Due to diagnostic uncertainty, 40% of HIV patients with fever and cough receive dual TB and histoplasmosis therapy. Their current standard of TB care includes sputum AFB microscopy and culture. However, rapid results are only available for the sputum AFB, which has a sensitivity of approximately 30%. The urine LAM Ag test is not presently used there. When combined with the urine LAM Ag test, sputum AFB has a sensitivity of 25% (if CD4>200) to 72% (if CD4<50). Over the next year, investigators plan to study changes in physician diagnostic classification and management decisions before and after the introduction of the urine LAM Ag test. This information would not only aid in TB diagnosis, but also in the investigators understanding of how physicians integrate new information.

The main objective is to determine the effect of urine LAM Ag test results in reducing dual TB/histoplasmosis therapy, by comparing the rate and duration of dual therapy in the urine LAM group to a retrospective control group. The investigators second objective is to investigate barriers to incorporating the urine LAM Ag test and how the results impact physicians' approaches to treatment using a physician questionnaire.

A clinical trial study will be conducted using HIV positive patients from June 2016 to June 2017 who present with pertinent clinical criteria at Hospital Santo Tomás. Following urine LAM Ag test administration, results will immediately be provided to the treating physicians. The control group will consist of retrospectively selected patients from the Hospital Santo Tomás database who fit the same inclusion and exclusion, matched for age, sex, and clinical severity. Patient outcome data will be collected from the day of hospital admittance to their time of discharge. Following the conclusion of data collection, consenting physicians will be interviewed on benefits and barriers to incorporating the urine LAM Ag test within their practice.

ELIGIBILITY:
Inclusion Criteria:

* HIV positive adult, and
* Admitted to Hospital Santo Tomas, and
* history of fevers, and
* Two or more of the following symptoms:

  * cough
  * shortness of breath
  * night sweats
  * weight loss
  * fatigue
  * loss of appetite

Exclusion Criteria:

* Under 18 yrs of age, or
* Already on TB therapy, or
* Anuric

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-11 (Estimated); Primary Completion 2018-08 (Estimated); Study Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
Dual therapy duration | 1 Week
  The number of days that anti-histoplasmosis and anti-tubercular medications are co-administered
Physician questionnaire | 1 year
  The questionnaire will be measured by Physician responses of Strongly Agree, Agree, Neutral, Disagree, or Strongly Disagree.

SECONDARY OUTCOMES:
Creatinine change during hospitalization | 1 week
  The change in baseline and peak creatinine levels during hospitalization
Number of diagnostic tests performed during hospitalization | 1 week
  Number of diagnostic tests performed during hospitalization
Mortality during hospital stay | 1 week
  Mortality during hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Amy Y Vittor, MD PHD, Principal Investigator — University of Florida

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Gutierrez ME, Canton A, Sosa N, Puga E, Talavera L. Disseminated histoplasmosis in patients with AIDS in Panama: a review of 104 cases. Clin Infect Dis. 2005 Apr 15;40(8):1199-202. doi: 10.1086/428842. Epub 2005 Mar 2. PMID 15791523
- [Background] Colombo AL, Tobon A, Restrepo A, Queiroz-Telles F, Nucci M. Epidemiology of endemic systemic fungal infections in Latin America. Med Mycol. 2011 Nov;49(8):785-98. doi: 10.3109/13693786.2011.577821. Epub 2011 May 4. PMID 21539506
- [Background] Vittor AY, Garland JM, Schlossberg D. Improving the diagnosis of tuberculosis: From QuantiFERON to new techniques to diagnose tuberculosis infections. Curr HIV/AIDS Rep. 2011 Sep;8(3):153-63. doi: 10.1007/s11904-011-0083-7. PMID 21660459
- [Background] Van Rie A, Page-Shipp L, Hanrahan CF, Schnippel K, Dansey H, Bassett J, Clouse K, Scott L, Stevens W, Sanne I. Point-of-care Xpert(R) MTB/RIF for smear-negative tuberculosis suspects at a primary care clinic in South Africa. Int J Tuberc Lung Dis. 2013 Mar;17(3):368-72. doi: 10.5588/ijtld.12.0392. PMID 23407225
- [Background] Lawn SD. Point-of-care detection of lipoarabinomannan (LAM) in urine for diagnosis of HIV-associated tuberculosis: a state of the art review. BMC Infect Dis. 2012 Apr 26;12:103. doi: 10.1186/1471-2334-12-103. PMID 22536883
- [Background] Wheat LJ, Connolly-Stringfield PA, Baker RL, Curfman MF, Eads ME, Israel KS, Norris SA, Webb DH, Zeckel ML. Disseminated histoplasmosis in the acquired immune deficiency syndrome: clinical findings, diagnosis and treatment, and review of the literature. Medicine (Baltimore). 1990 Nov;69(6):361-74. doi: 10.1097/00005792-199011000-00004. PMID 2233233
- [Background] Laurence YV, Griffiths UK, Vassall A. Costs to Health Services and the Patient of Treating Tuberculosis: A Systematic Literature Review. Pharmacoeconomics. 2015 Sep;33(9):939-55. doi: 10.1007/s40273-015-0279-6. PMID 25939501
- [Background] Rudolf F, Joaquim LC, Vieira C, Bjerregaard-Andersen M, Andersen A, Erlandsen M, Sodemann M, Andersen PL, Wejse C. The Bandim tuberculosis score: reliability and comparison with the Karnofsky performance score. Scand J Infect Dis. 2013 Apr;45(4):256-64. doi: 10.3109/00365548.2012.731077. Epub 2012 Oct 31. PMID 23113626